CLINICAL TRIAL: NCT01373671
Title: Multi-center Case Collection Study to Create a Library of Images From Various Approved FFDM Systems and 3D Images From Siemens Inspiration Digital Breast Tomosynthesis (DBT) System for Studies in Support of the Inspiration DBT Approval
Brief Title: Evaluation of the Efficacy of Digital Breast Tomosynthesis Imaging
Acronym: DBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siemens Medical Solutions USA - CSG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SMS-SP09-01
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: Mammography; Screening; Diagnostic
MeSH Terms: conditions — Breast Neoplasms; Disease | interventions — Mammography; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mammography exam (Other): Siemens DBT scan
  Interventions: Device: SIEMENS INSPIRATION DIGITAL BREAST TOMOSYNTHESIS (DBT) SYSTEM

INTERVENTIONS:
Device: SIEMENS INSPIRATION DIGITAL BREAST TOMOSYNTHESIS (DBT) SYSTEM — DBT scan

SUMMARY:
The primary objective of this protocol is to collect the 2-dimensional (2D) screening and diagnostic images, and 3-dimensional (3D) Digital Breast Tomosynthesis (DBT) scans from patient mammography examinations acquired on various commercially available Full Field Digital Mammography (FFDM) systems and the Siemens Inspiration DBT system, respectively.

DETAILED DESCRIPTION:
The image collection includes FFDM images and both raw and presentation data from the DBT system. The FFDM mammograms are performed using standard care screening or diagnostic mammography from various commercially available FFDM systems. All DBT images are acquired on the Inspiration DBT system specifically for the study, in addition to the clinically indicated screening mammograms. DBT images are read at the clinical sites and any DBT findings were investigated according to standard care.

ELIGIBILITY:
Inclusion Criteria:

All subjects enrolled into the collection study must:

* Provide signed informed consent after receiving a verbal and written explanation of the purpose and nature of the study
* be females, 40 years of age or older at the screening mammographic evaluation or age 30 or older presenting for a biopsy and have one of the following mammograms:

  o Normal cases at screening (BI-RADS® 1, 2 and 3):
  * have a screening mammogram that includes the four standard screening views (RCC, RMLO, LCC and LMLO), as well as have both MLO and CC DBT scans of each breast,

    o Actionable cases at screening (BI-RADS® 0, 4 or 5) with final BI-RADS® 1, 2, 3, 4 or 5:
  * have a screening mammogram with four SSVs and any clinically necessary diagnostic mammographic views, such as straight lateral projections, rolled, magnification view and spot compression views, and, both MLO and CC DBT scans of each breast plus 4 SSVs repeated at the diagnostic or biopsy visit if the screening images are unavailable or were acquired more than 45 days prior to DBT acquisition,
* have supporting ground-truth documentation for the final BI-RADS® assessment as follows:

  * A one (1) year FFDM follow up without evidence of cancer for normal cases not undergoing biopsy
  * A six (6) or twelve (12) month FFDM follow up confirming benign status for biopsy proven benign cases
  * Pathology report for either benign or malignant biopsy finding

Exclusion Criteria:

Subjects with any of the following conditions or who have had the following procedures will be excluded from this study:

* Pregnant women or women who believe they may be pregnant or are trying to become pregnant.
* Mastectomy patients
* Subjects who have had lumpectomy ≤ 5 years prior to the study entry
* Inmates (in accordance with 45 CFR 46.306) or mentally disabled individuals
* BI-RADS® Category 6 (e.g., for which the mammogram was performed for the purpose of planning cancer therapy)
* BI-RADS® Category 4 or 5 without confirming pathology reports will be considered incomplete
* Subjects with mammograms that lack the required views or with views judged to be technically inadequate will be considered incomplete and the cases will not be considered for the MRMC reader studies
* Subjects being accrued from the screening population who know that they will not be in the United States or available for follow up mammograms in one year.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 764 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Lazar — Siemens Medical Solutions USA, Inc
Locations (1):
- Siemens Medical Solutions, Malvern, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mammography Exam
Started | 764
Completed | 672
Not Completed | 92

BASELINE CHARACTERISTICS:
Arm/Group | Mammography Exam
Number analyzed (Participants) | 764
Age, Customized [Number; unit: participants] — >= 40 years >= 30 years if presenting for biopsy
  participants
    >= 40 years old | 752
    >= 30 years old < 40 | 12
Sex/Gender, Customized [Count of Participants; unit: Participants] — Female
  Participants
    Female | 764
Region of Enrollment [Number; unit: participants]
  United States | 764

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Based on the Area Under the Receiver Operating Characteristic (ROC) Curve in Breasts Analyzed With DBT as an Adjunct to FFDM vs. FFDM Alone
Description: The primary objective of this study was to demonstrate the superiority of DBT and FFDM images together in comparison to FFDM images alone with respect to the ability of readers to detect and diagnose malignant lesions. A comparison of the breast-level ROC areas was used to evaluate the superiority of DBT as an adjunct to FFDM vs. FFDM alone.
Time Frame: 1 year
Population: Per protocol 300 subjects were selected for analysis based on 89% power & 5% type one error rate determination.
Measure: Mean (Standard Error); unit: unitless
Units Other Than Participants: breasts
Groups:
- FFDM and DBT: FFDM exam and DBT scan on Siemens MAMMOMAT Inspiration
- FFDM Only: FFDM exam only
Arm/Group | FFDM and DBT | FFDM Only
Number analyzed (Participants) | 300 | 300
Number analyzed (breasts) | 490 | 490
unitless | 0.8527 (0.0268) | 0.7516 (0.0281)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Mammography Exam
Serious Adverse Events (participants affected / at risk) | 2/764
Other Adverse Events (participants affected / at risk) | 1/764
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mammography Exam (N=764)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 — Subject passed away from pneumonia. The SAE was not device related. Assessed around 1 year follow up.
Ovarian cancer (Reproductive system and breast disorders) | 1 — Subject passed away from ovarian cancer. The SAE was not device related. Assessed around time of 1 year follow up.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mammography Exam (N=764)
Lightheadedness (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less